CLINICAL TRIAL: NCT01113047
Title: An Open-label, Multicenter Study to Evaluate the Efficacy and Safety of a 4 Week Therapy With the Single Pill (SPC) Combination of Aliskiren 300 mg / Amlodipine 10 mg in Hypertensive Patients Not Adequately Respond to an Uptitrated 4 Week Therapy With the SPC of Olmesartan 40 mg / Amlodipine 10 mg, With a Potential Extension if Patients Still Not Adequately Respond With a 4 Week Therapy With the SPC Aliskiren 300 mg / Amlodipine 10 mg / HCTZ 12,5 mg
Brief Title: Aliskiren in Combination With Amlodipine in Hypertensive Patients Not Responding to Angiotensin Receptor Blocker (ARB) Plus Amlodipine
Acronym: AWESOME
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPA100ADE01
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Essential Hypertension
Keywords: Hypertension; Aliskiren; Amlodipine
MeSH Terms: conditions — Essential Hypertension; Hypertension | interventions — aliskiren; Amlodipine

ARMS (1):
- Non responder Olmesartan/Amlodipine (Experimental): Aliskiren/Amlodipine and Aliskiren/Amlodipine/HCTZ
  Interventions: Drug: Aliskiren/Amlodipine and Aliskiren/Amlodipine/HCTZ

INTERVENTIONS:
Drug: Aliskiren/Amlodipine and Aliskiren/Amlodipine/HCTZ — Aliskiren 300 mg / Amlodipine 10 mg/HCTZ 12.5 mg

SUMMARY:
This study will assess the efficacy and safety of the single pill combination of Aliskiren and Amlodipine in patients with moderate hypertension not adequately responding to a single pill combination of Olmesartan and Amlodipine.

Further this study will also assess the efficacy and safety of a single pill combination of Aliskiren, Amlodipine and Hydrochlorothiazide (HCTZ) in patients with moderate hypertension not adequately responding to a single pill combination of Aliskiren and Amlodipine.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension stage II
* Male and female patients
* Age >= 18 years old

Exclusion Criteria:

* Severe hypertension (systolic BP >= 180 mmHg, diastolic BP >= 110 mmHg
* Poorly controlled diabetes mellitus or type 1 DM
* History of myocardial infarction, stroke
* Presence of heart failure
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in mean sitting diastolic blood pressure after 4 weeks of treatment | 4 weeks

SECONDARY OUTCOMES:
Change in mean sitting systolic blood pressure reduction after 4 weeks of treatment with Aliskiren/Amlodipine or after 4 weeks of treatment with Aliskiren/Amlodipine/HCT | 4 weeks
Change in mean sitting diastolic blood pressure after 4 weeks of treatment with Aliskiren/Amlodipine/HCT | 4 weeks
Change in heart rate, pulse pressure, responder rates, normalization rates after 4 weeks of treatment with Aliskiren/Amlodipine or after 4 weeks of treatment with Aliskiren/Amlodipine/HCT | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Axthelm, Dr. med., Study Director — Novartis Pharmaceuticals
Locations (1):
- Investigative Site, Pirna, Germany

REFERENCES:
- [Derived] Axthelm C, Sieder C, Meister F, Pittrow D, Kaiser E. Aliskiren/amlodipine as a single-pill combination in hypertensive patients: subgroup analysis of elderly patients, with metabolic risk factors or high body mass index. J Drug Assess. 2012 Dec 25;2(1):1-10. doi: 10.3109/21556660.2012.762367. eCollection 2013. PMID 27536431